CLINICAL TRIAL: NCT00677352
Title: A Randomized, Double-Blind, Multicenter Study Of Sertraline Compared With Paroxetine In The Treatment Of Panic Disorder
Brief Title: A Study Of Sertraline Compared With Paroxetine In The Treatment Of Panic Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0501088
Record Dates: First submitted 2008-05-09; First posted 2008-05-14 (Estimated); Results first posted 2011-05-06 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Panic Disorder
Keywords: Panic Disorder
MeSH Terms: conditions — Panic Disorder | interventions — Sertraline; Paroxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: sertraline
- 2 (Active Comparator)
  Interventions: Drug: Paroxetine

INTERVENTIONS:
Drug: sertraline — dosage : 25mg , 50mg , placebo; dosage form : tablet; frequency : once daily after dinner; duration : 14 weeks
  Other Names: Zoloft, JZoloft
  Arms: 1
Drug: Paroxetine — dosage : 10mg, placebo; dosage form : capsule; frequency : once daily after dinner; duration : 14 weeks
  Other Names: Paxil
  Arms: 2

SUMMARY:
To evaluate the efficacy and safety of sertraline compared to paroxetine in patients with panic disorder.

ELIGIBILITY:
Inclusion Criteria:

* Patient who meets diagnosis of Panic Disorder (with or without Agoraphobia) according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM IV).
* Patients must have experienced at least 4 panic attacks within 4 weeks before screening.
* At baseline patients with Panic Disorder of total score of 18 or higher on the Panic and Agoraphobia scale (clinician rated version).

Exclusion Criteria:

* Patients who concurrently have bipolar disorder, schizophrenia, delusional disorder, epilepsy, Major Depression Disorder (MDD), Obsessive Compulsive Disorder (OCD), Seasonal Affective Disorder (SAD) or General Anxiety Disorder (GAD) according to the DSM-IV criteria.
* Patients who concurrently have depression/depressive state, anxiety disorder and generalized anxiety disorder may be included in the study if the primary diagnosis is identified to be panic disorder
* Patients with the total score of at least 18 on the Hamilton Depression Rating Scale (HAM-D) (Items 1 to 17) at the start of Screening (Visit 1)
* Patients who require concomitant drug therapy with psychotropic agents (including benzodiazepines) and monoamine oxidase inhibitor during the period of the study.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 321 (Actual)
Dates: Start 2008-05; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- Japan (22):
  - Pfizer Investigational Site, Nagoya, Aichi-ken
  - Pfizer Investigational Site, Fukuoka, Fukuoka
  - Pfizer Investigational Site, Kitakyushu-shi, Fukuoka
  - Pfizer Investigational Site, Kitakyusyu-shi, Fukuoka
  - Pfizer Investigational Site, Sapporo, Hokkaido
  - Pfizer Investigational Site, Higashiibaraki-gun, Ibaraki
  - Pfizer Investigational Site, Fujisawa, Kanagawa
  - Pfizer Investigational Site, Sagamihara-Shi, Kanagawa
  - Pfizer Investigational Site, Yokohama, Kanagawa
  - Pfizer Investigational Site, Kawaguchi-shi, Saitama
  - Pfizer Investigational Site, Saitama, Saitama
  - Pfizer Investigational Site, Chiyoda-ku, Tokyo
  - Pfizer Investigational Site, Kita-ku, Tokyo
  - Pfizer Investigational Site, Minato-ku, Tokyo
  - Pfizer Investigational Site, Musashino, Tokyo
  - Pfizer Investigational Site, Nakano-Ku, Tokyo
  - Pfizer Investigational Site, Nakanoku, Tokyo
  - Pfizer Investigational Site, Setagaya-ku, Tokyo
  - Pfizer Investigational Site, Shinjuku-ku, Tokyo
  - Pfizer Investigational Site, Toshima-ku, Tokyo
  - Pfizer Investigational Site, Nakano, Yokohama
  - Pfizer Investigational Site, Minatoku

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0501088&StudyName=A%20Study%20Of%20Sertraline%20Compared%20With%20Paroxetine%20In%20The%20Treatment%20Of%20Panic%20Disorder

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened at 34 centers in Japan.
Pre-assignment Details: Subjects who experienced at least one panic attack that met the DSM-IV diagnostic criteria per week between the start of the washout/observation period and the start of the double-blind treatment period and who had a total score of 18 or higher on the Panic and Agoraphobia Scale at the start of the double-blind treatment period.
Groups:
- Sertraline: Treatment phase was started from 25 mg/day followed by increase to 50 mg/day at Week 1, and treatment was continued for 3 weeks. If there was no tolerability concern at Week 4 at the discretion of the investigator (or subinvestigator), the dose was increased to 75 mg/day and treatment was continued for 2 weeks. If there was no tolerability concern at Week 6 at the discretion of the investigator (or subinvestigator), the dose was increased to 100 mg/day.
  At tapering phase, 50 mg/day was administered for 1 week after Week 12, followed by 25 mg/day for 1 week, and no study medication during the last 2 weeks.
- Paroxetine: Treatment phase was started from 10 mg/day followed by increase to 20 mg/day at Week 1, and treatment was continued for 3 weeks. If there was no tolerability concern at Week 4 at the discretion of the investigator (or subinvestigator), the dose was increased to 30 mg/day and treatment was continued for 2 weeks. If there was no tolerability concern at Week 6 at the discretion of the investigator (or subinvestigator), the dose was increased to 30 mg/day.
  At tapering phase, 20 mg/day was administered for 1 week after Week 12, followed by 10 mg/day for 1 week, and no study medication during the last 2 weeks.
Period: Treatment Phase
Arm/Group | Sertraline | Paroxetine
Started | 157 (All 157 subjects were treated with Sertraline.) | 164 (2 subjects were not teated, therefore 162 subjects were treated with paroxetine.)
Completed | 132 | 122
Not Completed | 25 | 42
Not completed — Adverse Event | 14 | 22
Not completed — Lack of Efficacy | 2 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 7 | 7
Not completed — Physician Decision | 1 | 0
Not completed — Pregnancy | 0 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Transference or work related matter | 0 | 5
Not completed — Not treated | 0 | 2
Period: Tapering Phase
Arm/Group | Sertraline | Paroxetine
Started | 132 | 122
Completed | 126 | 112
Not Completed | 6 | 10
Not completed — Adverse Event | 1 | 5
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Pregnancy | 0 | 1
Not completed — Job transfer | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sertraline | Paroxetine | Total
Number analyzed (Participants) | 157 | 162 | 319
Age, Customized [Number; unit: participants]
  < 18 years | 0 | 0 | 0
  18 - 44 years | 119 | 126 | 245
  45 -64 years | 38 | 36 | 74
  >= 65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 109 | 222
  Male | 44 | 53 | 97

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Panic and Agoraphobia Scale (PAS) Total Score at the End of Treatment Phase
Description: Panic and Agoraphobia Scale has 13 items with a 5-point scale (range: 0 to 4). The total possible score is ranged from 0 to 52. The increasing value are considered worse outcome. The scale is grouped into 5 subscores (not including item U in total score): panic attacks ; agoraphobia/avoidance behavior ; anticipatory anxiety; disability; and health worries. Four point difference in reduction of the PAS total score has been identified as not clinically meaningful in the assessment of Panic Disorder symptomatology.
Time Frame: Baseline and 12 weeks
Population: Efficacy Evaluable Set: A subset of patients in the Full Analysis Set who met some inclusion (diagnosis of Panic Disorder, etc.) and exclusion (psychotherapy, etc.) criteria, had to be treated for a minimum of 8 weeks and had a PAS score at least one evaluation during Week 8 to 12.
  Last Observation Carried Forward
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on scale
Arm/Group | Sertraline | Paroxetine
Number analyzed (Participants) | 127 | 127
Scores on scale | -17.4 [-18.9 to -15.9] | -17.0 [-18.4 to -15.5]
Statistical Analysis 1: Comparison: Sertraline vs Paroxetine; The two-sided 95% confidence interval (CI) of the intergroup difference (sertraline group - paroxetine group) of the mean reduction in the PAS total score at each dose during the treatment phase was calculated using an analysis of covariance (ANCOVA) model with treatment group as a factor and baseline PAS total score as a covariate; Test type: Non-Inferiority or Equivalence — Sertraline was concluded to be non-inferior to paroxetine when the upper limit of the CI fell below the non-inferiority margin of 4; ANCOVA; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-2.5 to 1.6]

2. Secondary Outcome: Percentage of Participants of Responder in Clinical Global Impression (CGI) - Improvement
Description: The ratings were rated to compare with baseline by 7-point " 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, 7 = very much worse".
  Responder was defined as number of participants who were assessed as "very much improved" or " much improved".
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Sertraline | Paroxetine
Number analyzed (Participants) | 127 | 127
Percentage of participants | 83.5 | 85.0

3. Secondary Outcome: Mean Change From Baseline in Panic Attack at the End of Treatment Phase
Description: Panic attacks were defined as having four or more of the following Diagnostic and Statistical Manual of Mental Disorders symptoms. Palpitations or increased heart rate, Sweating, Trembling or shaking, Shortness of breath or smothering sensations, Choking, Chest pain or discomfort, Nausea or upset stomach, Dizziness, unsteady feelings or faintness, Feeling unlike yourself, or detached from a situation and/or like things happening around you are strange and unreal, Fear of going crazy or doing something uncontrolled, Fear of dying, Abnormal sense, Hot flashes or chills.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: panic attacks per week
Arm/Group | Sertraline | Paroxetine
Number analyzed (Participants) | 127 | 127
panic attacks per week | -4.07 (6.12) | -4.59 (7.52)

4. Secondary Outcome: Mean Change From Baseline in Hamilton Anxiety Rating Scale Total Score at the End of Treatment Phase
Description: The Hamilton Anxiety Rating Scale provided a 5-point intensity rating (0=None to 4=Very severe) of anxiety symptoms in 14 items.
  The increasing values are considered worse outcome. The total possible score is ranged from 0 to 52.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sertraline | Paroxetine
Number analyzed (Participants) | 127 | 127
Scores on a scale | -11.35 (10.45) | -10.36 (8.27)

5. Secondary Outcome: Number of Participants With Summary of Adverse Events in Treatment Phase
Description: Number of sparticipants with all causality adverse events, serious adverse events, severe adverse events, adverse events resulted in discontinuation, dose reduced or temporary discontinuation. Participants were counted only once per treatment in each row.
Time Frame: 1, 2, 4, 6, 8 10 and 12 weeks (or study discontinuation) after administration of study drug
Population: The safety analysis set : Subset of patients who had taken at least one dose of the study drug and who had visited the study center at least once after taking the study drug.
Measure: Number; unit: Participants
Arm/Group | Sertraline | Paroxetine
Number analyzed (Participants) | 157 | 162
Participants
  Subjects with adverse events | 127 | 134
  Subjects with serious adverse events | 1 | 1
  Subjects with severe adverse events | 3 | 14
  Subjects discontinued due to adverse events | 14 | 23
  Dose reduced or temporary discontinuation | 13 | 14

6. Secondary Outcome: Summary of Adverse Events in Tapering Phase
Description: Number of subjects with all causality adverse events, serious adverse events, severe adverse events, adverse events resulted in discontinuation, dose reduced or temporary discontinuation. Subjects were counted only once per treatment in each row.
Time Frame: 4 weeks
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Sertraline | Paroxetine
Number analyzed (Participants) | 132 | 122
Participants
  Subjects with adverse events | 73 | 87
  Subjects with serious adverse events | 1 | 0
  Subjects with severe adverse events | 11 | 16
  Subjects discontinued due to adverse events | 1 | 4
  Dose reduced or temporary discontinuation | 0 | 0

7. Secondary Outcome: Percentage of Participants With Deterioration in Antidepressant Discontinuation Scale During Tapering Phase
Description: The percentage of participants divided was calcurated as follows: Devide the number of participants who had experienced new symptoms in Week 16, regardless of causal relationship with the study drug, or worsening of the severity in Week 16 compared with Week 12, by total number of participants in each treatment group.
Time Frame: 4 weeks
Population: Completer Set : Subset of patients in the EES who had a PAS rating at Week 16.
Measure: Number; unit: Percentage of participants
Arm/Group | Sertraline | Paroxetine
Number analyzed (Participants) | 124 | 118
Percentage of participants | 59.7 | 76.3
Statistical Analysis 1: Comparison: Sertraline vs Paroxetine; Test type: Superiority or Other; p = 0.0062, Fisher Exact — The p-value is not adjusted for multiple comparisons. A priori threshold for statistical significance is 0.05 (two-sided)

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Sertraline | Paroxetine
Serious Adverse Events (participants affected / at risk) | 2/157 | 1/162
Other Adverse Events (participants affected / at risk) | 132/157 | 137/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sertraline (N=157) | Paroxetine (N=162)
Enteritis infectious (Infections and infestations) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sertraline (N=157) | Paroxetine (N=162)
Palpitations (Cardiac disorders) | 7 | 10
Tachycardia (Cardiac disorders) | 5 | 13
Tinnitus (Ear and labyrinth disorders) | 1 | 10
Vertigo (Ear and labyrinth disorders) | 7 | 21
Abdominal discomfort (Gastrointestinal disorders) | 7 | 6
Abdominal pain upper (Gastrointestinal disorders) | 11 | 8
Constipation (Gastrointestinal disorders) | 7 | 23
Diarrhoea (Gastrointestinal disorders) | 37 | 29
Dry mouth (Gastrointestinal disorders) | 15 | 10
Nausea (Gastrointestinal disorders) | 43 | 66
Stomatitis (Gastrointestinal disorders) | 5 | 1
Vomiting (Gastrointestinal disorders) | 7 | 13
Asthenia (General disorders) | 7 | 15
Chills (General disorders) | 9 | 16
Fatigue (General disorders) | 12 | 17
Feeling jittery (General disorders) | 6 | 15
Irritability (General disorders) | 8 | 22
Malaise (General disorders) | 12 | 17
Thirst (General disorders) | 6 | 7
Nasopharyngitis (Infections and infestations) | 37 | 35
Decreased appetite (Metabolism and nutrition disorders) | 6 | 9
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 7 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 16
Disturbance in attention (Nervous system disorders) | 9 | 19
Dizziness (Nervous system disorders) | 42 | 61
Headache (Nervous system disorders) | 20 | 47
Hypoaesthesia (Nervous system disorders) | 5 | 9
Myoclonus (Nervous system disorders) | 4 | 6
Paraesthesia (Nervous system disorders) | 4 | 11
Somnolence (Nervous system disorders) | 34 | 62
Tremor (Nervous system disorders) | 6 | 19
Abnormal dreams (Psychiatric disorders) | 4 | 11
Anxiety (Psychiatric disorders) | 16 | 24
Depression (Psychiatric disorders) | 9 | 14
Insomnia (Psychiatric disorders) | 19 | 30
Mood altered (Psychiatric disorders) | 8 | 15
Panic disorder (Psychiatric disorders) | 2 | 6
Yawning (Respiratory, thoracic and mediastinal disorders) | 3 | 8
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 16 | 18
Urticaria (Skin and subcutaneous tissue disorders) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.